CLINICAL TRIAL: NCT03873116
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate the Efficacy and Safety of Two Dose Levels of BCX7353 as an Oral Treatment for the Prevention of Attacks in Subjects With Hereditary Angioedema
Brief Title: Study to Evaluate the Efficacy and Safety of BCX7353 as an Oral Treatment for the Prevention of HAE Attacks in Japan
Acronym: APeX-J
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioCryst Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: BCX7353-301
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Results first posted 2021-03-04 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-02

CONDITIONS: Hereditary Angioedema, HAE
Keywords: BCX7353
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — berotralstat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BCX7353 110mg once daily (Experimental): BCX7353 capsules administered orally once daily
  Interventions: Drug: BCX7353 capsules
- BCX7353 150mg once daily (Experimental): BCX7353 capsules administered orally once daily
  Interventions: Drug: BCX7353 capsules
- Placebo (Placebo Comparator): Matching placebo oral capsules administered orally once daily
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: BCX7353 capsules — BCX7353 capsules administered orally once daily
  Arms: BCX7353 110mg once daily
Drug: BCX7353 capsules — BCX7353 capsules administered orally once daily
  Arms: BCX7353 150mg once daily
Drug: Placebo oral capsule — Matching placebo capsules administered orally once daily
  Arms: Placebo

SUMMARY:
This is a phase 3, multi-center, randomized, double-blind, placebo-controlled trial to evaluate the efficacy and safety of oral BCX7353 in preventing acute angioedema attacks in patients with Type I and Type II HAE who live in Japan.

ELIGIBILITY:
Key Inclusion Criteria:

* A clinical diagnosis of hereditary angioedema (HAE) Type 1 or Type 2, defined as having a C1-INH functional level and a C4 level below the lower limit of the normal (LLN) reference range, as assessed during the Screening period.
* Access to and ability to use one or more acute medications approved by the relevant competent authority for the treatment of acute attacks of HAE
* Subjects must be medically appropriate for on-demand treatment as the sole medicinal management for their HAE during the study.
* Subjects must have a specified number of expert-confirmed attacks during the run-in period of 56 days from the Screening visit.
* Acceptable effective contraception
* Written informed consent

Key Exclusion Criteria:

* Pregnancy or breast-feeding
* Any clinically significant medical condition or medical history that, in the opinion of the Investigator or Sponsor, would interfere with the subject's safety or ability to participate in the study
* Any laboratory parameter abnormality that, in the opinion of the Investigator, is clinically significant and relevant for this study
* Severe hypersensitivity to multiple medicinal products or severe hypersensitivity/ anaphylaxis with unclear etiology
* Use of C1-INH within 14 days or use of androgens or tranexamic acid within 28 days prior to the Screening visit for prophylaxis of HAE attacks, or initiation of these drugs during the study
* Current participation in any other investigational drug study or received another investigational drug within 30 days of the Screening visit
* Prior enrollment in a BCX7353 study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-12-27 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isao Ohsawa, Principal Investigator — Saiyu Soka Hospital
Locations (10):
- Japan (10):
  - Study Site, Chiba
  - Study Site, Gunma
  - Study Site, Hokkaido
  - Study Site, Nagoya
  - Study Site, Osaka
  - Study Center, Saga
  - Study Site, Saitama
  - Study Site, Shimane
  - Study Site, Shizuoka
  - Study Site, Tokyo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Honda D, Hide M, Fukuda T, Koga K, Morita E, Moriwaki S, Sasaki Y, Suzuki Y, Collis P, Johnston DT, Tomita D, Desai B, Ohsawa I. Berotralstat for long-term prophylaxis of hereditary angioedema in Japan: Parts 2 and 3 of the randomized APeX-J Phase III trial. World Allergy Organ J. 2024 Mar 2;17(3):100882. doi: 10.1016/j.waojou.2024.100882. eCollection 2024 Mar. PMID 38445295
- [Derived] Farkas H, Balla Z. A review of berotralstat for the treatment of hereditary angioedema. Expert Rev Clin Immunol. 2023 Feb;19(2):145-153. doi: 10.1080/1744666X.2023.2150611. Epub 2022 Nov 29. PMID 36408587
- [Derived] Beard N, Frese M, Smertina E, Mere P, Katelaris C, Mills K. Interventions for the long-term prevention of hereditary angioedema attacks. Cochrane Database Syst Rev. 2022 Nov 3;11(11):CD013403. doi: 10.1002/14651858.CD013403.pub2. PMID 36326435
- [Derived] Ohsawa I, Honda D, Suzuki Y, Fukuda T, Kohga K, Morita E, Moriwaki S, Ishikawa O, Sasaki Y, Tago M, Chittick G, Cornpropst M, Murray SC, Dobo SM, Nagy E, Van Dyke S, Reese L, Best JM, Iocca H, Collis P, Sheridan WP, Hide M. Oral berotralstat for the prophylaxis of hereditary angioedema attacks in patients in Japan: A phase 3 randomized trial. Allergy. 2021 Jun;76(6):1789-1799. doi: 10.1111/all.14670. Epub 2020 Dec 23. PMID 33247955

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects with HAE Type 1 or Type 2 were eligible for the study following assessment of data obtained from screening procedures, including demonstration of a minimum number of qualifying angioedema events documented during a prospective run-in period of 56 days from the date of the screening visit. Randomization was stratified by the angioedema event rate over the period between screening and randomization (≥ 2 angioedema events per month vs. < 2 angioedema events per month).
Groups:
- Berotralstat 110mg Once Daily: Berotralstat administered as two 55mg capsules, orally QD in parts 1, 2 & 3.
- Berotralstat 110mg QD, Followed by Berotralstat 150 mg QD: Subjects were treated with 110 mg berotralstat QD in part 1 & 2 (up to 52 weeks) & 150 mg berotralstat QD in part 3 (52-104 weeks).
- Berotralstat 110mg QD After Placebo: Subjects were treated with placebo for 24 weeks in Part 1 and 110 mg berotralstat QD in part 2 (24-52 weeks) & part 3 (52-104 weeks).
- Berotralstat 110mg QD, Followed by Berotralstat 150 mg QD, After Placebo: Subjects were treated with placebo for 24 weeks in Part 1, 110 mg berotralstat QD in part 2 (24-52 weeks) & 150 mg berotralstat QD in part 3 (52-104 weeks).
- Berotralstat 150mg Once Daily: Berotralstat administered as two 75mg capsules, orally QD in parts 1, 2 & 3.
- Berotralstat 150mg QD After Placebo: Subjects were treated with placebo for 24 weeks in Part 1 and 150 mg berotralstat QD in part 2 (24-52 weeks) & part 3 (52-104 weeks).
Period: Part 1
Arm/Group | Berotralstat 110mg Once Daily | Berotralstat 110mg QD, Followed by Berotralstat 150 mg QD | Berotralstat 110mg QD After Placebo | Berotralstat 110mg QD, Followed by Berotralstat 150 mg QD, After Placebo | Berotralstat 150mg Once Daily | Berotralstat 150mg QD After Placebo
Started | 3 | 3 | 2 | 1 | 7 | 3
Completed | 3 | 3 | 2 | 1 | 7 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Study drug discontinuation due to rash | 0 | 0 | 0 | 0 | 0 | 1
Period: Part 2
Arm/Group | Berotralstat 110mg Once Daily | Berotralstat 110mg QD, Followed by Berotralstat 150 mg QD | Berotralstat 110mg QD After Placebo | Berotralstat 110mg QD, Followed by Berotralstat 150 mg QD, After Placebo | Berotralstat 150mg Once Daily | Berotralstat 150mg QD After Placebo
Started | 3 | 3 | 1 (One subject receiving Placebo in Part 1, withdrew from the study before part 2.) | 1 | 7 | 2
Completed | 3 | 3 | 0 | 1 | 6 | 2
Not Completed | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lab abnormality or AE | 0 | 0 | 0 | 0 | 1 | 0
Period: Part 3
Arm/Group | Berotralstat 110mg Once Daily | Berotralstat 110mg QD, Followed by Berotralstat 150 mg QD | Berotralstat 110mg QD After Placebo | Berotralstat 110mg QD, Followed by Berotralstat 150 mg QD, After Placebo | Berotralstat 150mg Once Daily | Berotralstat 150mg QD After Placebo
Started | 0 (Three Subjects withdrew consent at week 52 visit - end part 2) | 3 | 0 | 1 | 6 | 1 (One Subject withdrew consent at week 52 visit - end part 2)
Completed | 0 | 3 | 0 | 1 | 5 | 1
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part 1: Berotralstat 110mg Once Daily: Berotralstat administered as two 55mg capsules, orally QD for 24 weeks.
- Part 1: Berotralstat 150mg Once Daily: Berotralstat administered as two 75mg capsules, orally QD for 24 weeks.
- Part 1: Placebo: Placebo administered as two 2 matching capsules, orally QD for24 weeks.
- Total: Total of all reporting groups
Arm/Group | Part 1: Berotralstat 110mg Once Daily | Part 1: Berotralstat 150mg Once Daily | Part 1: Placebo | Total
Number analyzed (Participants) | 6 | 7 | 6 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (15.03) | 37.3 (9.05) | 42.3 (13.52) | 42.1 (12.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 5 | 16
  Male | 1 | 1 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 6 | 6 | 6 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Baseline expert-confirmed angioedema event rate [Number; unit: participants]
  ≥ 2 events/month | 2 | 4 | 3 | 9
  < 2 events/month | 4 | 3 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Part 1: The Rate of Expert-confirmed HAE Attacks During Dosing in the Entire 24-week Treatment Period (Day 1 to Day 168)
Description: The angioedema event rate and the treatment comparisons between each berotralstat dose and placebo in the rate of expert-confirmed angioedema events during the entire dosing period was analyzed using a negative binomial regression model. The number of expert-confirmed angioedema events was included as the dependent variable, the treatment was included as a fixed effect, the stratification variable (baseline monthly angioedema event rate) and study (for the combined study analysis) were included as covariates, and the logarithm of duration on treatment was included as an offset variable. The estimated rate of angioedema events for each treatment group, the treatment differences expressed as the angioedema event rate ratio (berotralstat) over placebo rate ratio), and their associated 95% confidence intervals (CIs) were provided from the negative binomial regression model.
Time Frame: 24 weeks
Population: The intent to treat (ITT) population included all randomized subjects, regardless of whether study treatment was administered. This population was the primary population for the analysis of the efficacy and health outcomes data.
Measure: Mean (Standard Deviation); unit: Angioedema event rate per 28 days
Groups:
- Berotralstat 110mg Once Daily: Berotralstat administered as two 55mg capsules, orally QD for 24 weeks.
- Berotralstat 150mg Once Daily: Berotralstat administered as two 75mg capsules, orally QD for 24 weeks.
- Placebo: Placebo administered as two matching capsules, orally QD for 24 weeks.
Arm/Group | Berotralstat 110mg Once Daily | Berotralstat 150mg Once Daily | Placebo
Number analyzed (Participants) | 6 | 7 | 6
Angioedema event rate per 28 days | 1.961 (1.3021) | 1.089 (0.9168) | 2.734 (1.6359)
Statistical Analysis 1: Comparison: Berotralstat 110mg Once Daily vs Placebo; Test type: Superiority; p = 0.181, negative binomial regression model; negative binomial regression model = -24.6, 95% CI 2-sided [-50.1 to 14.0]
Statistical Analysis 2: Comparison: Berotralstat 150mg Once Daily vs Placebo; Test type: Superiority; p = 0.003, negative binomial regression model; negative binomial regression model = -49.1, 95% CI 2-sided [-67.5 to -20.4]

2. Primary Outcome: Part 2: To Evaluate the Long-term Safety and Tolerability of Berotralstat 110 and 150 mg in Subjects With HAE
Description: The safety data was assessed for the safety population for subjects who entered Part 2, and includes TEAEs that occurred in Part 1 and Part 2 for these subjects with a data cut-off date of 10-April-2020. TEAEs are defined as AEs that occurred on or after first dose of study treatment, whether in Part 1 or 2, and were assigned to the relevant treatment depending on when the TEAE began (Part 1 or Part 2 treatment). TEAEs were assessed for severity (graded) using the Division of Microbiology and Infectious Disease (DMID) criteria for grading AEs. TEAEs not covered by the DMID criteria were assessed as Mild (Grade 1), Moderate (Grade 2), Severe (Grade 3) or Life-threatening (Grade 4).
Time Frame: Part 1: 24 weeks (Week 0 to 24 to 52), Part 2: 28 weeks (Week 24 to 52)
Population: The safety population included all subjects who received at least 1 capsule of study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Berotralstat 110mg Once Daily: Berotralstat administered as two 55mg capsules, orally QD in parts 1 & 2.
- Berotralstat 110mg QD After Placebo: Subjects were treated with 110 mg berotralstat QD in part 2 (24-52 weeks), following part 1 placebo treatment.
- Berotralstat 150mg Once Daily: Berotralstat administered as two 75mg capsules, orally QD in parts 1 & 2.
- Berotralstat 150mg QD After Placebo: Subjects were treated with 150 mg berotralstat QD in part 2 (24-52 weeks), following part 1 placebo treatment.
- Placebo: Subjects were treated with Placebo in Part 1
Arm/Group | Berotralstat 110mg Once Daily | Berotralstat 110mg QD After Placebo | Berotralstat 150mg Once Daily | Berotralstat 150mg QD After Placebo | Placebo
Number analyzed (Participants) | 6 | 2 | 7 | 2 | 6
Participants
  TEAE | 6 | 1 | 7 | 2 | 6
  Drug-related TEAE | 2 | 0 | 3 | 0 | 2
  SAE | 2 | 0 | 0 | 0 | 0
  Drug-related SAE | 0 | 0 | 0 | 0 | 0
  Grade 3 or 4 TEAE | 0 | 0 | 1 | 0 | 1
  Drug-related grade 3 or 4 TEAE | 0 | 0 | 1 | 0 | 0
  TEAE leading to interruption of study drug | 1 | 0 | 2 | 0 | 0
  TEAE leading to discontinuation of study drug | 0 | 0 | 1 | 0 | 1
  Investigator-identified rash (event of special interest) | 1 | 0 | 2 | 0 | 1
  GI abdominal related TEAE | 3 | 1 | 3 | 1 | 1
  GI abdominal related TEAE leading to discontinuation of study drug | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Part 3: To Evaluate the Long-term Safety and Tolerability of Berotralstat Administered QD Over a 52- to up to 104-week Administration Period in Subjects With HAE.
Description: The safety data was assessed for the safety population for subjects who entered Part 3, and includes TEAEs that occurred in Part 3 for these subjects.
Time Frame: Part 3: Week 52 to up to Week 104.
Measure: Count of Participants; unit: Participants
Groups:
- Berotralstat 150mg Once Daily: Berotralstat administered as two 75mg capsules, orally QD.
Arm/Group | Berotralstat 150mg Once Daily
Number analyzed (Participants) | 11
Participants
  TEAE | 6
  Drug-related TEAE | 0
  SAE | 1
  Drug-related SAE | 0
  Grade 3 or 4 TEAE | 1
  Drug-related grade 3 or 4 TEAE | 0
  TEAE leading to interruption of study drug | 0
  TEAE leading to discontinuation of study drug | 0
  Investigator-identified rash (event of special interest) | 0
  GI abdominal related TEAE | 0
  GI abdominal related TEAE leading to discontinuation of study drug | 0

4. Secondary Outcome: Part 1: Proportion of Days With Angioedema Symptoms Through 24 Weeks.
Description: Assessment of number and proportion of days subjects had angioedema symptoms from expert-confirmed angioedema events during Part 1.
Time Frame: 24 weeks
Population: The ITT population included all randomized subjects, regardless of whether study treatment was administered. This population was the primary population for the analysis of the efficacy and health outcomes data. Data were analyzed according to randomized treatment.
Measure: Least Squares Mean (Standard Error); unit: Proportion days with angioedema symptoms
Arm/Group | Berotralstat 110mg Once Daily | Berotralstat 150mg Once Daily | Placebo
Number analyzed (Participants) | 6 | 7 | 6
Proportion days with angioedema symptoms | 0.258 (0.0534) | 0.118 (0.0500) | 0.240 (0.0536)
Statistical Analysis 1: Comparison: Berotralstat 110mg Once Daily vs Placebo; Numerical differences from the placebo treatment in the LSM proportion of the 169 days of treatment with angioedema symptoms; Test type: Superiority; p = 0.814, ANCOVA; Difference in Least Square Means = 0.018, 95% CI 2-sided [-0.143 to 0.179]
Statistical Analysis 2: Comparison: Berotralstat 150mg Once Daily vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.120, ANCOVA; Difference in Least Square Means = -0.122, 95% CI 2-sided [-0.280 to 0.036]

5. Secondary Outcome: Part 1: Rate of Expert-confirmed Angioedema Events During Dosing in the Effective Treatment Period
Description: The rate of expert-confirmed angioedema events for the effective treatment period gives an analysis of the efficacy of active treatment after berotralstat had reached steady-state concentrations, given the effective half-life of 150 mg berotralstat in Study BCX7353-106 (Study 106) of 89 hours.
Time Frame: Day 8 through to 24 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Angioedema event rate per 28 days
Arm/Group | Berotralstat 110mg Once Daily | Berotralstat 150mg Once Daily | Placebo
Number analyzed (Participants) | 6 | 7 | 6
Angioedema event rate per 28 days | 1.988 (1.3422) | 1.136 (0.9564) | 2.775 (1.6472)
Statistical Analysis 1: Comparison: Berotralstat 110mg Once Daily vs Placebo; In the event that the first secondary endpoint did not meet statistical significance in the hierarchical testing scheme, testing of the second secondary endpoint of rate of expert-confirmed angioedema events during dosing in the effective treatment period for statistical significance would not be completed. Therefore, P-values reported are nominal; Test type: Superiority; p = 0.188, mixed-model repeated measures analysis; mixed-model repeated measures analysis = 24.5, 95% CI 2-sided [-14.7 to 50.3]
Statistical Analysis 2: Comparison: Berotralstat 150mg Once Daily vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.005, mixed-model repeated measures analysis; mixed-model repeated measures analysis = 47.6, 95% CI 2-sided [17.7 to 66.6]

6. Secondary Outcome: Part 1: Change From Baseline in Angioedema Quality of Life (AE-QoL) Questionnaire at Week 24 (Total Score)
Description: Change in Quality of Life, on a 1-100 scale, where higher scores indicate more impairment and a decrease (change with a negative value) in AE-QoL questionnaire scores indicates an improvement in the subject's QoL. The minimum clinically important difference (MCID) for the AE-QoL questionnaire is -6 (total score).
Time Frame: Baseline and 24 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: AE-QoL Total Score Change from baseline
Arm/Group | Berotralstat 110mg Once Daily | Berotralstat 150mg Once Daily | Placebo
Number analyzed (Participants) | 6 | 7 | 6
AE-QoL Total Score Change from baseline | -9.47 (6.933) | -15.82 (6.424) | 3.18 (6.832)
Statistical Analysis 1: Comparison: Berotralstat 110mg Once Daily vs Placebo; Numerical difference in change from baseline of AE-QoL total score between treatment groups. In the event that the first secondary endpoint did not meet statistical significance in the hierarchical testing scheme, testing of the third secondary endpoint of change from baseline in AE-QoL total score at Week 24 for statistical significance would not be completed. P-values that are reported are nominal; Test type: Superiority; p = 0.213, mixed-model repeated measures analysis; mixed-model repeated measures analysis = -12.65, 95% CI 2-sided [-33.33 to 8.03]
Statistical Analysis 2: Comparison: Berotralstat 150mg Once Daily vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.061, mixed-model repeated measures analysis; mixed-model repeated measures analysis = -19.00, 95% CI 2-sided [-39.00 to 0.99]

7. Secondary Outcome: Part 2: To Assess the Effectiveness of Berotralstat Over a 24- to 52-week Period
Description: Monthly Attack Rate was defined as the total number of investigator-confirmed HAE attacks experienced during the treatment period adjusted for the length of a month (defined as 28 days) and the number of days the subject was on treatment during that month. The end of Month 6 was defined as the start of Part 2 treatment. For crossover subjects receiving active treatment following placebo, months were adjusted according to the date of the first dose of active treatment.
  Baseline investigator-confirmed attack rate was defined as the total number of investigator-confirmed HAE attacks experienced in the period between screening and first dose of study drug adjusted for the length of a month (defined as 28 days) and the number of days during that period.
Time Frame: 28 weeks (Week 24 to 52)
Population: The intent to treat (ITT) population included all randomized subjects, regardless of whether study treatment was administered. This population was the primary population for the analysis of the efficacy data.
Measure: Mean (Standard Deviation); unit: HAE attacks/28 days-change from baseline
Arm/Group | Berotralstat 110mg Once Daily | Berotralstat 110mg QD After Placebo | Berotralstat 150mg Once Daily | Berotralstat 150mg QD After Placebo
Number analyzed (Participants) | 6 | 2 | 7 | 2
HAE attacks/28 days-change from baseline
  Month 6 | -0.487 (1.0661) | -0.686 (0.2872) | -0.863 (1.3000) | -1.386 (0.5951)
  Month 7: number analyzed (Participants) | 6 | 1 | 7 | 2
  Month 7 | -1.085 (0.8249) | -0.889 (0) | -1.395 (0.9127) | -1.403 (0.7948)
  Month 8: number analyzed (Participants) | 6 | 0 | 7 | 0
  Month 8 | -0.585 (0.5622) |  | -1.395 (0.8016) |
  Month 9: number analyzed (Participants) | 6 | 0 | 7 | 0
  Month 9 | -0.418 (0.8910) |  | -0.927 (0.7645) |
  Month 10: number analyzed (Participants) | 6 | 0 | 6 | 0
  Month 10 | -0.918 (1.0134) |  | -0.733 (0.8068) |
  Month 11: number analyzed (Participants) | 6 | 0 | 6 | 0
  Month 11 | -0.585 (0.5622) |  | -1.400 (0.9997) |
  Month 12: number analyzed (Participants) | 6 | 0 | 6 | 0
  Month 12 | -0.585 (1.0737) |  | -0.900 (0.3925) |
  Month 13: number analyzed (Participants) | 6 | 0 | 6 | 0
  Month 13 | -0.757 (0.9729) |  | -0.733 (1.3060) |

8. Secondary Outcome: Part 2: To Evaluate QoL Following Berotralstat Administration Over a 24- to 52-week Period.
Description: Change in Quality of Life, on a 1-100 scale, where higher scores indicate more impairment and a decrease (change with a negative value) in AE-QoL questionnaire scores indicates an improvement in the subject's QoL. The minimum clinically important difference (MCID) for the AE-QoL questionnaire is -6 (total score). The AE-QoL is only validated for adults; however, data were collected on all adult and adolescent study subjects.
Time Frame: 28 Weeks (Week 24 to 52)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: AE-QoL score -change from baseline
Arm/Group | Berotralstat 110mg Once Daily | Berotralstat 110mg QD After Placebo | Berotralstat 150mg Once Daily | Berotralstat 150mg QD After Placebo
Number analyzed (Participants) | 6 | 1 | 7 | 1
AE-QoL score -change from baseline
  Week 24 | -4.9 (13.0) | -19.1 (0) | -19.5 (31.2) | 0 (0)
  Week 52: number analyzed (Participants) | 4 | 0 | 7 | 0
  Week 52 | -7.4 (9.4) |  | -17.2 (30.6) |

9. Secondary Outcome: Part 3: To Assess the Effectiveness of Berotralstat Over a 52- to up to 104-week Administration Period
Description: Adjusted subject-reported event rate was defined as (total number of adjusted subject-reported HAE events experienced in the period between the Week 52 visit and end of study [or the last dose date/time in Part 3 + 24 hours for subjects who discontinued drug in Part 3]) * 28/(date of last dose in Part 3 - date of Week 52 visit + 1).
Time Frame: 52 weeks (Week 52 to 104)
Population: The intent to treat (ITT) population included all randomized subjects, regardless of whether study treatment was administered. This population was the primary population for the analysis of the efficacy data. The rate of adjusted subject-reported events for subjects treated in Part 3 is presented.
Measure: Mean (Standard Deviation); unit: HAE attacks per 28 days
Arm/Group | Berotralstat 150mg Once Daily
Number analyzed (Participants) | 11
HAE attacks per 28 days | 0.883 (1.1216)

10. Secondary Outcome: Part 3: To Evaluate QoL Following Berotralstat Administration Over a 52- to up to 104-week Period
Description: Change in Quality of Life, on a 1-100 scale, where higher scores indicate more impairment and a decrease (change with a negative value) in AE-QoL questionnaire scores indicates an improvement in the subject's QoL. The minimum clinically important difference (MCID) for the AE-QoL questionnaire is -6 (total score). For subjects who received active treatment following placebo, visits were adjusted according to the date of the first dose of active treatment.
Time Frame: 52 Weeks (Week 52 to 104)
Population: The intent to treat (ITT) population included all randomized subjects, regardless of whether study treatment was administered. This population was the primary population for the analysis of the efficacy data. QoL for subjects treated in Part 3 is presented.
Measure: Mean (Standard Deviation); unit: AE-QoL score -change from baseline
Groups:
- Berotralstat 150mg Once Daily: Berotralstat administered as two 75mg capsules, orally QD during part 3
Arm/Group | Berotralstat 150mg Once Daily
Number analyzed (Participants) | 11
AE-QoL score -change from baseline
  Week 52: number analyzed (Participants) | 9
  Week 52 | -11.11 (29.089)
  Week 60 | -13.24 (23.758)
  Week 72 | -17.38 (24.998)
  Week 84 | -11.63 (22.900)
  Week 96: number analyzed (Participants) | 8
  Week 96 | -20.40 (32.069)
  Week 104: number analyzed (Participants) | 8
  Week 104 | -18.93 (30.681)

11. Secondary Outcome: Part 3: To Evaluate Subject's Satisfaction With Berotralstat During 52- to 104-week Administration Period
Description: The Treatment Satisfaction Questionnaire for Medication (TSQM) was completed by subjects at baseline and at each study visit until the end of the study. TSQM scores consisted of 14 items of which 13 items were made up of 3 specific scales (Effectiveness, Side Effects, and Convenience) and 1 global satisfaction scale (Global Satisfaction). At baseline, TSQM questionnaires were completed based on subject's satisfaction with usual medications. At all other time points for collection of TSQM, subjects were asked about their level of satisfaction or dissatisfaction with the study drug. Scales scores were calculated for each scale and were transformed into scores ranging from 0 to 100, with higher scores indicating higher satisfaction. TSQM score and corresponding change from baseline values were calculated at each visit. For subjects who received active treatment following placebo, visits were adjusted according to the date of the first dose of active treatment.
Time Frame: 52 Weeks (Week 52 to 104)
Population: The intent to treat (ITT) population included all randomized subjects, regardless of whether study treatment was administered. This population was the primary population for the analysis of the efficacy data. TSQM global scores for subjects treated in Part 3 is presented.
Measure: Mean (Standard Deviation); unit: TSQM Global score -change from baseline
Groups:
- Berotralstat 150mg Once Daily: Berotralstat administered orally as two 75mg capsules (150 mg QD) or two 50 mg capsules (100 mg QD).
Arm/Group | Berotralstat 150mg Once Daily
Number analyzed (Participants) | 11
TSQM Global score -change from baseline
  Week 60 | 11.7 (37.15)
  Week 72 | 13.6 (37.72)
  Week 84 | 11.7 (34.44)
  Week 96: number analyzed (Participants) | 8
  Week 96 | 18.8 (26.43)
  Week 104: number analyzed (Participants) | 8
  Week 104 | 16.1 (23.77)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were assessed and recorded from the time that the Informed consent form was signed until the last follow-up visit, approximately 3 weeks following the last dose of study drug, or until the AE was resolved or the subject was in a clinically stable condition with regard to the AE. AEs were assigned to the relevant treatment depending on when the AE began; i.e., Part 1 or Part 2 and 3 treatment.
Groups:
- Berotralstat 110mg Once Daily: Berotralstat administered as two 55mg capsules, orally QD
- Placebo: Placebo administered as two matching capsules, orally QD
Arm/Group | Berotralstat 110mg Once Daily | Berotralstat 150mg Once Daily | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/9 | 0/6
Serious Adverse Events (participants affected / at risk) | 2/8 | 1/9 | 0/6
Other Adverse Events (participants affected / at risk) | 8/8 | 9/9 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Berotralstat 110mg Once Daily (N=8) | Berotralstat 150mg Once Daily (N=9) | Placebo (N=6)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hereditary angioedema (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Berotralstat 110mg Once Daily (N=8) | Berotralstat 150mg Once Daily (N=9) | Placebo (N=6)
Nasopharyngitis (Infections and infestations) | 3 (3) | 4 (4) | 4 (5)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (5) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (8) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophageal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 1 (92) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (2) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vaccination site joint swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertrigliceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-08-07): https://cdn.clinicaltrials.gov/large-docs/16/NCT03873116/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-04): https://cdn.clinicaltrials.gov/large-docs/16/NCT03873116/SAP_001.pdf